CLINICAL TRIAL: NCT02106143
Title: A Prospective Study of RejuvenAir™ System Radial Spray Cryotherapy to Determine Safety and Histological Effect in the Lung
Brief Title: RejuvenAir™ System Lobectomy Safety and Histology Study
Acronym: Lobectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CSA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 009
Record Dates: First submitted 2014-04-02; First posted 2014-04-08 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Lung Neoplasms; Airway Obstruction; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Airway Obstruction

STUDY DESIGN:
Intervention Model Description: RejuvenAir
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RejuvenAir™ Radial Spray Cryotherapy (Experimental): Subjects will receive Rejuvenair Radial SCT prior to lobectomy.
  Interventions: Device: RejuvenAir™ Radial Spray Cryotherapy

INTERVENTIONS:
Device: RejuvenAir™ Radial Spray Cryotherapy — Metered dose radial spray cryotherapy treatment

SUMMARY:
Cryotherapy has a long history of safe use in various medical procedures. RejuvenAir System radial spray cryotherapy is a novel procedure being developed as a treatment for conditions associated with abnormal bronchial function, such as chronic bronchitis. The development of appropriate reliable equipment, definition of therapeutic parameters, and an understanding of the tissue effects of treatment have been established through animal studies. This clinical study is being undertaken to assess the feasibility and safety of the application of a radial metered dose spray cryotherapy in the human airway and to evaluate the treatment depth in human airways. The study design is prospective, open label, single arm multi-center study that will consist of up to 15 subjects at up to 3 enrolling sites in Ireland, UK and The Netherlands RejuvenAir System treatment will be performed during preoperative bronchoscopy 0 to 60 days prior to prescheduled lung resection in Subjects requiring lobectomy or pneumonectomy for removal of peripheral tumors. Treatment will be limited to areas of the bronchi within the lobe that will be removed, distal to the anticipated margin of resection. Treatment should be at least 1 cm from the bronchial resection margins and away from the tumor bed. Treated airways will be inspected via bronchoscopy at the time of thoracotomy, and examined histologically following surgical resection. Subject participation will be from 1 to 60 days and enrollment is anticipated to take 4-5 months.Total study duration is expected to last approximately 10 months.

DETAILED DESCRIPTION:
The patient population intended to participate in this study are subjects scheduled to undergo lobectomy/pneomonectomy for peripheral lung lesions suspicious for or known to be cancer. The intention is that the spray cryotherapy dosing will be performed at the same surgical session as the intended surgery. Bronchoscopy is routinely performed just prior to the start of the lung resection and it is anticipated that the spray cryotherapy dose will be delivered at that time. Care will be taken to avoid administration of the spray cryotherapy dose at or near the surgical resection margin or near the lung lesion itself.

A secondary endpoint beyond the safety and ease of delivery of the spray cryotherapy dose will be an analysis of the local tissue effect of the spray cryotherapy dose. Given that this area will reside within the anticipated resected surgical specimen, the treatment site will be inspected for evidence of depth of tissue effect using routine hematoxylin and eosin staining and light microscopy evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of 21 to 75 years of age.
* Subject is able to read, understand, and sign a written Informed Consent to participate in the study.
* Subject is scheduled within 60 days, for a total lobectomy or pneumonectomy procedure unrelated to this study (upper and lower lobes only).
* Subject has a pre-procedure post bronchodilator FEV1 of greater than or equal to 50% of predicted.
* Subject is able to undergo bronchoscopy in the opinion of the investigator or per hospital guidelines.
* Subject is able to adhere to and undergo a scheduled bronchoscope procedure prior to their clinically scheduled lobectomy or pneumonectomy surgical procedure.

Exclusion Criteria:

* Subject is pregnant, nursing, or planning to get pregnant during study duration.
* Subject has had prior radiation therapy which involved the lungs.
* Subject has received chemotherapy within the past 6 months, or is anticipated to be treated with chemotherapy between initial study treatment and lobectomy/pneumonectomy procedure.
* Subject has an acute pulmonary infection or pneumonia within 6 weeks prior to study bronchoscopy.
* Subject has had COPD exacerbation within 6 weeks prior to study bronchoscopy.
* Subject has bronchiectasis in the area to be treated.
* Subject has bullous emphysema. Characterized as large bullae >3 centimeters and confirmed on CT.
* Subject has had a transplant.
* Subject has had lung reduction surgery, including emphysema stent (s) implanted, coils or other devices for emphysema implanted.
* Subject has uncontrolled coagulopathy or bleeding disorder.
* Subject has participated in another clinical study within 6 weeks of baseline.
* Subject has a serious medical condition, such as: uncontrolled congestive heart failure, uncontrolled angina, myocardial infarction in the past year, renal failure, liver disease, cerebrovascular accident within the past 6 months, uncontrolled diabetes, hypertension, autoimmune disease or uncontrolled gastric reflux.
* Subject has known sensitivity to medication required to perform bronchoscopy (such as lidocaine, atropine, and benzodiazepines).

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
safety | 2 months
  Safety as measured by occurrence of serious adverse events related to metered dose radial spray cryotherapy treatment performed prior to scheduled lobectomy or pneumonectomy surgery

SECONDARY OUTCOMES:
Measurement of histological changes at treatment sites | 2 months
  Description of depth of histological treatment effect per specified treatment dose

CONTACTS AND LOCATIONS:
Overall Officials: David Breen, MD, Study Chair — Galway University Hospital; Pallav Shah, MD, Study Chair — Royal Brompton & Harefield NHS Foundation Trust; Dirk-Jan Slebos, MD, Study Chair — University Medical Center Geoningen
Locations (3):
- Galway University Hosptial, Galway, Galway, Ireland
- University Medical Center Groningen, Groningen, Netherlands
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Au JT, Carson J, Monette S, Finley DJ. Spray cryotherapy is effective for bronchoscopic, endoscopic and open ablation of thoracic tissues. Interact Cardiovasc Thorac Surg. 2012 Oct;15(4):580-4. doi: 10.1093/icvts/ivs192. Epub 2012 Jul 18. PMID 22811511
- [Background] Krimsky WS, Broussard JN, Sarkar SA, Harley DP. Bronchoscopic spray cryotherapy: assessment of safety and depth of airway injury. J Thorac Cardiovasc Surg. 2010 Mar;139(3):781-2. doi: 10.1016/j.jtcvs.2009.03.051. Epub 2009 Aug 6. No abstract available. PMID 19664781
- [Background] Fernando HC, Dekeratry D, Downie G, Finley D, Sullivan V, Sarkar S, Rivas R Jr, Santos RS. Feasibility of spray cryotherapy and balloon dilation for non-malignant strictures of the airway. Eur J Cardiothorac Surg. 2011 Nov;40(5):1177-80. doi: 10.1016/j.ejcts.2011.02.062. Epub 2011 Apr 8. PMID 21482131
- [Background] Finley DJ, Dycoco J, Sarkar S, Krimsky WS, Sherwood JT, Dekeratry D, Downie G, Atwood J, Fernando HC, Rusch VW. Airway spray cryotherapy: initial outcomes from a multiinstitutional registry. Ann Thorac Surg. 2012 Jul;94(1):199-203; discussion 203-4. doi: 10.1016/j.athoracsur.2012.01.112. Epub 2012 Apr 18. PMID 22516831
- [Background] Krimsky WS, Rodrigues MP, Malayaman N, Sarkar S. Spray cryotherapy for the treatment of glottic and subglottic stenosis. Laryngoscope. 2010 Mar;120(3):473-7. doi: 10.1002/lary.20794. PMID 20058314
- [Background] Browning R, Parrish S, Sarkar S, Turner JF Jr. First report of a novel liquid nitrogen adjustable flow spray cryotherapy (SCT) device in the bronchoscopic treatment of disease of the central tracheo-bronchial airways. J Thorac Dis. 2013 Jun;5(3):E103-6. doi: 10.3978/j.issn.2072-1439.2013.05.26. No abstract available. PMID 23825781